CLINICAL TRIAL: NCT04255433
Title: The Effect of Tirzepatide Versus Dulaglutide on Major Adverse Cardiovascular Events in Patients With Type 2 Diabetes (SURPASS-CVOT)
Brief Title: A Study of Tirzepatide (LY3298176) Compared With Dulaglutide on Major Cardiovascular Events in Participants With Type 2 Diabetes
Acronym: SURPASS-CVOT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17073; I8F-MC-GPGN (Other: Eli Lilly and Company); 2019-002735-28 (EudraCT Number)
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Hypoglycemic Agents; Physiological Effects of Drugs; Tirzepatide; Incretins; Glucagon-Like Peptide 1; Gastric Inhibitory Polypeptide; Hormones; Hormones, Hormone Substitutes, and Hormone Antagonists
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases | interventions — Tirzepatide; dulaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tirzepatide (Experimental): Tirzepatide administered subcutaneously (SC) once a week.
  Interventions: Drug: Tirzepatide
- Dulaglutide (Active Comparator): Dulaglutide administered SC once a week.
  Interventions: Drug: Dulaglutide

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: Tirzepatide
Drug: Dulaglutide — Administered SC
  Other Names: LY2189265
  Arms: Dulaglutide

SUMMARY:
The purpose of the trial is to assess the efficacy and safety of tirzepatide to dulaglutide in participants with type 2 diabetes and increased cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 40 years old with a diagnosis of type 2 diabetes
* Established cardiovascular disease, including at least 1 of the following:

  * Coronary artery disease (CAD) with any of the following:

    * Documented history of spontaneous myocardial infarction (MI)
    * ≥50% stenosis in 1 or more major coronary arteries, determined by invasive angiography
    * ≥50% stenosis in 2 or more major coronary arteries, determined by computed tomography coronary angiography (CTCA)
    * History of surgical or percutaneous coronary revascularization procedure
  * Cerebrovascular disease - any of the following:

    * Documented history of ischemic stroke
    * Carotid arterial disease with ≥50% stenosis, documented by carotid ultrasound, magnetic resonance imaging (MRI), or angiography
    * Carotid stenting or surgical revascularization
  * Peripheral arterial disease with either of the following:

    * Intermittent claudication and ankle-brachial index <0.9
    * Prior nontraumatic amputation or peripheral vascular procedure (eg, stenting or surgical revascularization), due to peripheral arterial ischemia
  * Note: Supporting medical documentation is required in all instances
* HbA1c ≥7% (≥53 mmol/mol) and ≤10.5% (≤91.3 mmol/mol) based on central laboratory assessment at screening
* Body mass index (BMI) ≥25 kg/m2
* At the time of signing the informed consent: Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical trials.

  * Male patients: Men, regardless of their fertility status, with nonpregnant women of childbearing potential (WOCBP) partners must agree to either remain abstinent (if this is their preferred and usual lifestyle) or use condoms, as well as 1 additional highly effective (less than 1% failure rate) method of contraception (such as combination oral contraceptives, implanted contraceptives, or intrauterine devices) or effective method of contraception (such as diaphragms with spermicide or cervical sponges) for the duration of the study and until their plasma concentrations are below the level that could result in a relevant potential exposure to a possible fetus, predicted to be 90 days following the last dose of study drug.

    * Men and their partners may choose to use a double-barrier method of contraception. (Barrier protection methods without concomitant use of a spermicide are not an effective or acceptable method of contraception. Thus, each barrier method must include use of a spermicide. It should be noted, however, that the use of male and female condoms as a double barrier method is not considered acceptable due to the high failure rate when these barrier methods are combined).
    * Periodic abstinence (eg, calendar, ovulation, symptothermal, or postovulation methods), declaration of abstinence just for the duration of a trial, and withdrawal are not acceptable methods of contraception.
  * Men with pregnant partners should use condoms during intercourse for the duration of the study and until the end of the estimated relevant potential exposure in WOCBP (90 days). Men should refrain from sperm donation for the duration of the study and until their plasma concentrations are below the level that could result in a relevant potential exposure to a possible fetus, predicted to be 90 days following the last dose of study drug. Men who are in exclusively same-sex relationships (as their preferred and usual lifestyle) are not required to use contraception.
  * Female patients: Women of childbearing potential who are abstinent (if this is complete abstinence, as their preferred and usual lifestyle) or in a same-sex relationship (as part of their preferred and usual lifestyle) must agree to either remain abstinent or stay in a same-sex relationship without sexual relationships with males. Periodic abstinence (eg, calendar, ovulation, symptothermal, or postovulation methods), declaration of abstinence just for the duration of a trial, and withdrawal are not acceptable methods of contraception. Otherwise, WOCBP participating must agree to use 2 forms of effective contraception, where at least 1 form is highly effective (less than 1% failure rate), for the entirety of the study. Contraception must continue following completion of study drug administration for the entirety of the study and for 30 days thereafter.

    * WOCBP participating must test negative for pregnancy prior to initiation of treatment as indicated by a negative serum pregnancy test at the screening visit followed by a negative urine pregnancy test within 24 hours prior to exposure.
    * Two forms of effective contraception, where at least 1 form is highly effective, (such as combination oral contraceptives, implanted contraceptives, or intrauterine devices) will be used. Effective contraception (such as male or female condoms with spermicide, diaphragms with spermicide, or cervical sponges) may be used as the second therapy. Barrier protection methods without concomitant use of a spermicide are not a reliable or acceptable method. Thus, each barrier method must include use of a spermicide (ie, condom with spermicide, diaphragm with spermicide, or female condom with spermicide). It should be noted that the use of male and female condoms as a double barrier method is not considered acceptable due to the high failure rate when these methods are combined.
  * Women not of childbearing potential may participate and include those who are:

    * infertile due to surgical sterilization (hysterectomy, bilateral oophorectomy, or tubal ligation), congenital anomaly such as mullerian agenesis, or
    * postmenopausal - defined as either: A woman at least 40 years of age with an intact uterus, not on hormone therapy, who has cessation of menses for at least 1 year without an alternative medical cause, AND a follicle-stimulating hormone >40 mIU/mL; or ii. A woman 55 or older not on hormone therapy, who has had at least 12 months of spontaneous amenorrhea; or A woman at least 55 years of age with a diagnosis of menopause prior to starting hormone replacement therapy.
* In the investigator's opinion, are well motivated, capable, and willing to:

  * learn how to self-inject treatment (tirzepatide or dulaglutide), as required for this protocol (visually impaired persons who are not able to perform the injections must have the assistance of a sighted individual trained to inject the study drug; persons with physical limitations who are not able to perform the injections must have the assistance of an individual trained to inject the study drug),
  * inject study drug weekly,
  * have a sufficient understanding of 1 of the provided languages of the country such that they will be able to complete the patient questionnaires, and
  * make themselves available for the duration of the study, and who will comply with the required study visits.
* Capable of giving signed informed consent

Exclusion Criteria:

* Have type 1 diabetes mellitus
* Have uncontrolled diabetes requiring immediate therapy (such as diabetic ketoacidosis) at screening or randomization, in the judgment of the physician
* Have had 1 or more events of severe hypoglycemia and/or 1 or more events of hypoglycemia unawareness within 6 months prior to screening
* Are currently planning treatment for diabetic retinopathy and/or macular edema.
* Have been hospitalized for congestive heart failure (CHF) within 2 months prior to screening
* Have chronic New York Heart Association Functional Classification IV CHF
* Are currently planning a coronary, carotid, or peripheral artery revascularization
* Had chronic or acute pancreatitis any time prior to screening, irrespective of etiology
* Have a known clinically significant gastric emptying abnormality such as severe gastroparesis or gastric outlet obstruction, or have undergone or currently planning any gastric bypass (bariatric) surgery or restrictive bariatric surgery
* Have acute or chronic hepatitis, signs or symptoms of any other liver disease, an alanine aminotransferase (ALT) level ≥3 times the upper limit of normal (ULN) for the reference range, as determined by the central laboratory (Note: Patients with nonalcoholic fatty liver disease are eligible to participate if their ALT level is <3 times the ULN for the reference range)
* Have known chronic severe renal failure (defined as a known estimated glomerular filtration rate (eGFR) <15 mL/minute/1.73 m2) or are on chronic dialysis
* Have evidence of a significant, uncontrolled endocrine abnormality (eg, thyrotoxicosis or adrenal crises)
* Have a family or personal history of multiple endocrine neoplasia type 2 (MEN2) or familial medullary thyroid carcinoma (MTC) or personal history of nonfamilial MTC
* Have a serum calcitonin level at screening of: (based on central laboratory results)

  * ≥20 ng/L at Visit 1, if eGFR ≥60 mL/min/1.73 m2, or
  * ≥35 ng/L at Visit 1, if eGFR <60 mL/min/1.73 m2
* Have a history of an active or untreated malignancy or are in remission from a clinically significant malignancy for less than 5 years. An exception for this criterion is basal or squamous cell skin cancer, in situ carcinomas of the cervix, or in situ prostate cancer
* Have a history of any other condition (such as known drug or alcohol abuse or psychiatric disorder) that, in the opinion of the investigator, may preclude the patient from following and completing the protocol
* Have had a transplanted organ (corneal transplants [keratoplasty] allowed) or awaiting an organ transplant
* Have any other condition (eg, hypersensitivity) that is a contraindication to any incretin or glucagon-like peptide-1 (GLP-1) receptor agonist (RA)
* Have had an MI, percutaneous coronary revascularization procedure, ischemic stroke, carotid stenting or surgical revascularization, nontraumatic amputation, or peripheral vascular procedure (eg, stenting or surgical revascularization) less than 60 days prior to screening
* Have had coronary artery bypass graft surgery less than 5 years prior to screening
* Have had a blood transfusion or severe blood loss within 90 days prior to screening or have known hematological conditions that may interfere with HbA1c measurement
* Treatment with GLP-1 RA or pramlintide, in a period of 3 months prior to Visit 1
* Discontinuation of GLP-1 RA or pramlintide, due to intolerability any time prior to Visit 1
* Are currently enrolled in any other clinical study involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study
* Have participated within the last 30 days in a clinical trial involving an investigational product. If the previous investigational product has a long half-life, 3 months or 5 half-lives (whichever is longer) should have passed
* Have previously completed or withdrawn from this study or randomized into any other study investigating tirzepatide

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13299 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Time to First Occurrence of Death from Cardiovascular (CV) Causes, Myocardial Infarction (MI), or Stroke (MACE-3) | Randomization up to Study Completion (Approximate Maximum 54 Months)
  Time to First Occurrence of a component event of MACE-3

SECONDARY OUTCOMES:
Time to Death from Any Cause | Randomization up to Study Completion (Approximate Maximum 54 Months)
  Time to Death from Any Cause
Time to CV Death | Randomization up to Study Completion (Approximate Maximum 54 Months)
  Time to CV Death
Time to First Occurrence of MI | Randomization up to Study Completion (Approximate Maximum 54 Months)
  Time to First Occurrence of MI
Time to First Occurrence of Stroke | Randomization up to Study Completion (Approximate Maximum 54 Months)
  Time to First Occurrence of Stroke
Time to First Occurrence of the Expanded Composite of CV Death, MI, Stroke, Coronary Revascularization, or Hospitalization for Unstable Angina | Randomization up to Study Completion (Approximate Maximum 54 Months)
  Time to First Occurrence of the Expanded Composite of CV Death, MI, Stroke, Coronary Revascularization, or Hospitalization for Unstable Angina
Cumulative Number of CV Deaths and Total (First and Recurrent) Heart Failure Events Requiring Hospitalization and/or Urgent Heart Failure Visits | End of Study (Approximate Maximum 54 Months)
  Cumulative Number of CV Deaths and Total (First and Recurrent) Heart Failure Events Requiring Hospitalization and/or Urgent Heart Failure Visits
Percentage of Participants with More than 10% Weight Loss | 36 Months
  Percentage of Participants with More than 10% Weight Loss
Change from Baseline in Body Weight | Baseline, End of Study (Approximate Maximum 54 Months)
  Change from Baseline in Body Weight
Change from Baseline in Hemoglobin A1c (HbA1c) | Baseline, End of Study (Approximate Maximum 54 Months)
  Change from Baseline in HbA1c
Change from Baseline in Urinary Albumin to Creatinine Ratio | Baseline, End of Study (Approximate Maximum 54 Months)
  Change from Baseline in Urinary Albumin to Creatinine Ratio
Change from Baseline in Blood Lipids | Baseline, End of Study (Approximate Maximum 54 Months)
  Change from Baseline in Blood Lipids (Total Cholesterol, Low-Density Lipoprotein Cholesterol, High-Density Lipoprotein Cholesterol, and Triglycerides)
Time to First Occurrence of Revascularization | Randomization up to Study Completion (Approximate Maximum 54 Months)
  Time to First Occurrence of Revascularization
Time to First Occurrence of Hospitalization Due to Unstable Angina | Randomization up to Study Completion (Approximate Maximum 54 Months)
  Time to First Occurrence of Hospitalization Due to Unstable Angina
Time to First Occurrence of New or Worsening Nephropathy | Randomization up to Study Completion (Approximate Maximum 54 Months)
  Time to First Occurrence of New or Worsening Nephropathy
Cumulative Number of Primary Composite Events of CV Death and Total (First and Recurrent) MI and/or Stroke | End of Study (Approximate Maximum 54 Months)
  Cumulative Number of Primary Composite Events of CV Death and Total (First and Recurrent) MI and/or Stroke

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (632):
- United States (121):
  - University of Alabama at Birmingham Medical Center, Birmingham, Alabama
  - John Muir Medical Center - Concord Campus, Concord, California
  - Valley Clinical Trials, Inc., Covina, California
  - AMCR Institute, Escondido, California
  - Valley Research, Fresno, California
  - NorCal Medical Research, Inc, Greenbrae, California
  - UCSD - Altman Clinical and Translational Research Institute (ACTRI), La Jolla, California
  - First Valley Medical Group, Lancaster, California
  - Monterey Endocrine & Diabetes Institute, Inc., Monterey, California
  - Riverside University Health System - Medical Center, Moreno Valley, California
  - Diabetes Associates Medical Group, Orange, California
  - Pasadena Clinical Research, Pasadena, California
  - LCGK Research, San Carlos, California
  - Norcal Endocrinology & Internal Medicine, San Ramon, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - CMR of Greater New Haven, LLC, Hamden, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Orlando Heart & Vascular Institute, LLC, Altamonte Springs, Florida
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Encore Medical Research, Hollywood, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Accel Research Sites - St. Pete-Largo Clinical Research Unit, Largo, Florida
  - Ocala Caridovascular Research, Ocala, Florida
  - Cardiology Partners Clinical Research Institute - Palm Beach Gardens, Palm Beach Gardens, Florida
  - Peace River Cardiovascular Center, Port Charlotte, Florida
  - Professional Health Care of Pinellas, St. Petersburg, Florida
  - Cardiology Partners Clinical Research Institute - Wellington, Wellington, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Kaiser Permanente - Dutluth, GA, Duluth, Georgia
  - NSC Research, Johns Creek, Georgia
  - Physicians Research Associates, Lawrenceville, Georgia
  - East Coast Institute for Research at The Jones Center, Macon, Georgia
  - Atlanta Heart Specialists, Tucker, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - VA Pacific Islands Health Care System, Honolulu, Hawaii
  - Elite Clinical Trials, Blackfoot, Idaho
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Northwest Heart Clinical Research, Arlington Heights, Illinois
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Clinical Investigation Specialists, Gurnee, Illinois
  - Central Illinois Diabetes and Clinical Research a Division of Prairie Education and Research Cooperative, Springfield, Illinois
  - University of Iowa, Iowa City, Iowa
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - The University of Kansas - Clinical Research Center, Fairway, Kansas
  - Cotton O'Neil Diabetes & Endocrinology, Topeka, Kansas
  - Cotton O'Neil Mulvane, Topeka, Kansas
  - Qualmedica Research, Bowling Green, Kentucky
  - L-MARC Research Center, Louisville, Kentucky
  - Qualmedica Research, LLC, Owensboro, Kentucky
  - Ascension Saint Agnes Heart Care, Baltimore, Maryland
  - MedStar Health Research Institute (MedStar Physician Based Research Network), Hyattsville, Maryland
  - MD Medical Research, Oxon Hill, Maryland
  - Endocrine and Metabolic Consultants, Rockville, Maryland
  - Brigham and Women's Hospital Diabetes Program, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - ActivMed Practices and Research, Methuen, Massachusetts
  - Infinity Medical Research, North Dartmouth, Massachusetts
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - St. John's Hospital, Edina, Minnesota
  - M Health Fairview St. John's Hospital, Maplewood, Minnesota
  - CentraCare Heart & Vascular Center, Saint Cloud, Minnesota
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Clinvest Research LLC, Springfield, Missouri
  - Mercy Research - Smith Glynn Callaway, Springfield, Missouri
  - Billings Clinic, Billings, Montana
  - Mercury Street Medical Group, PLLC, Butte, Montana
  - VA Nebraska-Western Iowa Health Care System, Omaha, Nebraska
  - University Of Nebraska Medical Center, Omaha, Nebraska
  - Palm Research Center Tenaya, Las Vegas, Nevada
  - Palm Research Center Sunset, Las Vegas, Nevada
  - Southern Nh Diabetes and Endocrinology, Nashua, New Hampshire
  - Albany Medical College, Division of Community Endocrinology, Albany, New York
  - Great Lakes Medical Research, LLC, Westfield, New York
  - Atrium Health - Department of Family Medicine Research, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - PMG Research Inc., d/b/a PMG of Piedmont Healthcare, Mooresville, North Carolina
  - Accellacare - Wilmington, Wilmington, North Carolina
  - Lillestol Research, Fargo, North Dakota
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Alliance for Multispecialty Research, LLC, Norman, Oklahoma
  - Heritage Valley Medical Group, Inc., Beaver, Pennsylvania
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - Decpa, Llc, Feasterville, Pennsylvania
  - Thomas Jefferson University - Clinical Research Institute, Philadelphia, Pennsylvania
  - Northeast Endocrine Metabolic Associates, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians, Preferred Clinical Research (Ofc 18), Pittsburgh, Pennsylvania
  - Cardiology Consultants of Philadelphia Yardley, Yardley, Pennsylvania
  - Ralph H. Johnson VA Medical Center, Charleston, South Carolina
  - Tribe Clinical Research, LLC, Greenville, South Carolina
  - Accellacare - Mt Pleasant, Mt. Pleasant, South Carolina
  - Monument Health Rapid City Hospital, Rapid City, South Dakota
  - Holston Medical Group, Bristol, Tennessee
  - PMG Research, Inc. d/b/a PMG Research of Knoxville, Knoxville, Tennessee
  - Endocrine Clinic, Memphis, Tennessee
  - Private Practice - Dr. Osvaldo A. Brusco, Corpus Christi, Texas
  - Dallas Diabetes Research Center, Dallas, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - Research Institute of Dallas, Dallas, Texas
  - Texas Health Physicians Group, Dallas, Texas
  - Galenos Research, Dallas, Texas
  - Academy of Diabetes, Thyroid and Endocrine, El Paso, Texas
  - Diabetes and Thyroid Center of Ft. Worth, Fort Worth, Texas
  - Northwest Houston Cardiology - Cypress, Houston, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - North Hills Family Medicine/North Hills Medical Research, North Richland Hills, Texas
  - Audie L Murphy VA Hospital, San Antonio, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Northwest Houston Heart Center, Tomball, Texas
  - Physicians' Research Options, Draper, Utah
  - Advanced Research Institute, Ogden, Utah
  - Alpine Medical Group, Salt Lake City, Utah
  - Kalo Clinical Research, West Valley City, Utah
  - Virginia Heart, Falls Church, Virginia
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - VA Puget Sound Health Care System, Seattle, Washington
  - Multicare Institute for Research and Innovation, Spokane, Washington
  - Central Washington Health Services Association d/b/a Confluence Health, Wenatchee, Washington
  - Clinical Investigation Specialists, Kenosha, Wisconsin
- Argentina (31):
  - Instituto de Investigaciones Clínicas Bahia Blanca, Bahía Blanca, Buenos Aires
  - Organizacion Medica de Investigacion, CABA, Buenos Aires
  - CEDIC, CABA, Buenos Aires
  - Stat Research S.A., Capital Federal, Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata, Mar del Plata, Buenos Aires
  - DIM Clínica Privada, Ramos Mejía, Buenos Aires
  - Go Centro Medico San Nicolás, San Nicolás de los Arroyos, Buenos Aires
  - Instituto de Investigaciones Clinicas Zarate, Zárate, Buenos Aires
  - Centro Médico Viamonte, Buenos Aires, Buenos Aires F.D.
  - Mautalen Salud e Investigación, Buenos Aires, Buenos Aires F.D.
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires, Buenos Aires F.D.
  - CEMEDIAB, C.a.b.a., Buenos Aires F.D.
  - Centro Medico Privado CEMAIC, Capital, Córdoba Province
  - Centro Medico Privado San Vicente Diabetes, Córdoba, Córdoba Province
  - Instituto Médico Catamarca IMEC, Rosario, Santa Fe Province
  - Instituto Médico Fundación Grupo Colaborativo Rosario Investigación y Prevención Medica, Rosario, Santa Fe Province
  - Instituto de Investigaciones Clinicas Rosario, Rosario, Santa Fe Province
  - Centro de Investigaciones Médicas Tucuman, SAN M. de Tucuman, Tucumán Province
  - Clínica Mayo de Urgencias Médicas Cruz Blanca S.R.L, San Miguel de Tucumán, Tucumán Province
  - Investigaciones Clínicas Tucumán, San Miguel de Tucumán, Tucumán Province
  - CEMEDIC, Buenos Aires
  - Glenny Corp, Buenos Aires
  - CIPREC, Buenos Aires
  - Asociación de Beneficencia Hospital Sirio Libanés, Buenos Aires
  - Centro Universitario de Investigación en Farmacologia Clínic, Corrientes
  - Instituto de Cardiología "Juana F. Cabral", Corrientes
  - CIDIM-Centro Integral de Diagnostico por Imagenes Marchegiani, Córdoba
  - Centro Diabetológico Dr. Waitman, Córdoba
  - Instituto Médico Alas, Salta
  - Sanatorio Norte, Santiago del Estero
- Australia (20):
  - The AIM Centre / Hunter Diabetes Centre, Merewether, New South Wales
  - Nepean Hospital, Penrith, New South Wales
  - University of Sydney - Charles Perkins Centre, Sydney, New South Wales
  - Illawarra Shoalhaven Local Health District, Wollongong, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Core Research Group, Brisbane, Queensland
  - Mater Misericordiae Limited, Brisbane, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - The Townsville Hospital, Townsville, Queensland
  - Nightingale Research, Adelaide, South Australia
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Southern Adelaide Diabetes & Endocrine Services, Oaklands Park, South Australia
  - Launceston General Hospital, Launceston, Tasmania
  - Box Hill Hospital, Box Hill, Victoria
  - Victorian Heart Hospital, Clayton, Victoria
  - Barwon Health, Geelong, Victoria
  - Austin Health - Repatriation Hospital, Heidelberg West, Victoria
  - School of Medicine, Fremantle Hospital, Fremantle, Western Australia
  - Advara HeartCare Joondalup, Joondalup, Western Australia
  - GenesisCare - Murdoch - Murdoch Drive, Murdoch, Western Australia
- Austria (6):
  - Medizinische Universität Graz, Graz, Styria
  - Uniklinikum Salzburg, Salzburg
  - Klinik Landstraße, Vienna
  - Zentrum für klinische Studien Dr Hanusch Gmbh, Vienna
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna
  - Klinik Hietzing, Vienna
- Belgium (14):
  - Imelda General Hospital, Bonheiden, Antwerpen
  - Algemeen Ziekenhuis klina, Brasschaat, Antwerpen
  - Antwerp University Hospital, Edegem, Antwerpen
  - Université Libre de Bruxelles - Hôpital Erasme, Brussels, Bruxelles-Capitale, Région de
  - UZ Brussel, Brussels, Bruxelles-Capitale, Région de
  - ZAS Jan Palfijn, Merksem, Flanders
  - AZORG Campus Aalst-Moorselbaan, Aalst, Oost-Vlaanderen
  - AZ Nikolaas, Sint-Niklaas, Oost-Vlaanderen
  - UZ Leuven, Leuven, Vlaams-Brabant
  - AZ Sint-Jan Brugge-Oostende AV, Bruges, West-Vlaanderen
  - AZ Groeninge Campus Kennedylaan, Kortrijk, West-Vlaanderen
  - Az Damiaan vzw, Ostend, West-Vlaanderen
  - AZ Delta vzw, Roeselare, West-Vlaanderen
  - Centre Hospitalier Universitaire de Liège - Domaine Universitaire du Sart Tilman, Liège
- Brazil (14):
  - Private Practice - Dr.Miguel N. Hissa, Fortaleza, Ceará
  - CEDOES, Vitória, Espírito Santo
  - Quanta Diagnóstico e Terapia, Curitiba, Paraná
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Instituto de Pesquisa clinica de Campinas, Campinas, São Paulo
  - Loema Instituto de Pesquisa Clinica, Campinas, São Paulo
  - CECIP - Centro de Estudos do Interior Paulista, Jaú, São Paulo
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - ISPEM - Instituto São José dos Campos em Pesquisas Médicas, São José dos Campos, São Paulo
  - Instituto de Pesquisa Clinica, São Paulo, São Paulo
  - CPCLIN, São Paulo, São Paulo
  - IBPClin - Instituto Brasil de Pesquisa Clínica, Rio de Janeiro
  - CPQuali Pesquisa Clínica, São Paulo
  - Hospital das Clinicas FMUSP, São Paulo
- Canada (29):
  - LMC Diabetes & Endocrinology, Calgary, Alberta
  - BC Diabetes Office, Vancouver, British Columbia
  - Dr. M.B. Jones Inc., Victoria, British Columbia
  - Winnipeg Clinic, Winnipeg, Manitoba
  - NSHA-QEII Health Sciences Centre-Dickson Bldg, Halifax, Nova Scotia
  - LMC Clinical Research Inc. (Barrie), Barrie, Ontario
  - LMC Diabetes & Endocrinology, Brampton, Ontario
  - Aggarwal and Associates Limited, Brampton, Ontario
  - Cambridge Cardiac Care Centre, Cambridge, Ontario
  - LMC Clinical Research Inc. (Thornhill), Concord, Ontario
  - Janik Research Corporation, Greater Sudbury, Ontario
  - Milestone Research Inc., London, Ontario
  - St. Joseph's Health Care, London, Ontario
  - North York Diagnostic and Cardiac Centre, North York, Ontario
  - LMC Clinical Research Inc. (Oakville), Oakville, Ontario
  - Private Practice - Dr. James Cha, Oshawa, Ontario
  - LMC Manna Research, Ottawa, Ontario
  - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - Bluewater Clinical Research Group Inc., Sarnia, Ontario
  - Diabetes Clinic, Smiths Falls, Ontario
  - Canadian Phase Onward, Toronto, Ontario
  - LMC Clinical Research Inc. (Bayview), Toronto, Ontario
  - Diabetes Heart Research Centre, Toronto, Ontario
  - Dr. Anil K. Gupta Medicine Professional Corporation, Toronto, Ontario
  - Viacar Recherche Clinique, Greenfield Park, Quebec
  - Centre de Recherche Clinique de Laval, Laval, Quebec
  - Manna Research, Lévis, Quebec
  - Clinique Sante Cardio MC, Montreal, Quebec
  - Diex Recherche Quebec, Québec
- China (23):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Lanzhou university second hospital, Lanzhou, Gansu
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - First Huai'an Hospital Affiliated to Nanjing Medical University, Huai'an, Jiangsu
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jiangxi Pingxiang People's Hospital, Pingxiang, Jiangxi
  - China-Japan Union Hospital, Changchun, Jilin
  - The People's Hospital of Liaoning Province, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Jinan Central Hospital, Jinan, Shandong
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
- Czechia (10):
  - MUDr. Alena Vachova, České Budějovice, Jihočeský kraj
  - MUDr. Tomas Edelsberger, Krnov, Moravskoslezský kraj
  - Interni a diabetologicka ordinace, s.r.o., Náchod, Náchod
  - Diabet2 s.r.o., diabetologicka a interni ambulance, Prague, Praha 1
  - ResTrial s.r.o., Prague, Praha 8
  - MUDr. Barbora Diepoltova, Praha 9 - Klanovice, Praha 9
  - Diacentrum Brandys n.L. s.r.o., Brandýs nad Labem, Praha-východ
  - Vseobecna fakultni nemocnice v Praze, Prague
  - MUDr. Michala Pelikanova s.r.o., Prague
  - Milan Kvapil s.r.o., Diabetologicka ambulance, Prague
- France (11):
  - CHU Bordeaux Haut-Leveque, Pessac, Aquitaine
  - Groupe Hospitalier Mutualiste Les Portes du Sud, Vénissieux, Auvergne-Rhône-Alpes
  - Hôtel-Dieu du Creusot - site Harfleur, Le Creusot, Bourgogne-Franche-Comté
  - Centre Hospitalier Universitaire Dijon Bourgogne - Hôpital François Mitterrand, Dijon, Côte-d'Or
  - CHU Rangueil, Toulouse, Haute-Garonne
  - Hôpital Nord Guillaume-et-René-Laennec / CHU de Nantes, Saint-Herblain, Loire-Atlantique
  - Centre Hospitalier Régional Universitaire de Nancy - Hôpitaux de Brabois, Vandœuvre-lès-Nancy, Lorraine
  - Assistance Publique Hôpitaux de Paris - Groupe Hospitalier 10e - Hôpital Lariboisière, Paris
  - Hôpital Bichat - Claude-Bernard, Paris
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes, Île-de-France Region
  - Groupe hospitalier Paris saint Joseph, Paris, Île-de-France Region
- Germany (47):
  - Gemeinschaftspraxis Dres. Jung, Deggingen, Baden-Wurttemberg
  - Marienhospital Stuttgart, Stuttgart, Baden-Wurttemberg
  - Gemeinschaftspraxis Prof. Dr. med. Stephan Jacob, Dr. med. Frohmut Jacob, Villingen-Schwenningen, Baden-Wurttemberg
  - Praxis Sauter & Sauter & Vorbach, Wangen, Baden-Wurttemberg
  - CIMS Studienzentrum Bamberg, Bamberg, Bavaria
  - Private Practice - Dr. Ilka Simon-Wagner, Lichtenfels, Bavaria
  - CDG Studienambulanz Hartard, München, Bavaria
  - ZKS Suedbrandenburg, Elsterwerda, Brandenburg
  - ZKS Dr. Lüdemann, Falkensee, Brandenburg
  - ClinPhenomics GmbH & Co KG, Frankfurt am Main, Hesse
  - MVZ im Altstadt-Carree Fulda GmbH, Fulda, Hesse
  - Diabetes Zentrum Dr. Tews, Gelnhausen, Hesse
  - Diabetologische Schwerpunktpraxis Marck Linn Pickel, Pohlheim, Hesse
  - Praxis Oedeme, Lüneburg, Lower Saxony
  - Praxis Dr. Veronika Wenzl-Bauer, Rehlingen, Lower Saxony
  - Herz - und Diabeteszentrum Nordrhein - Westfalen, Bad Oeynhausen, Bad Oeynhausen, North Rhine-Westphalia
  - Diabetes- und Stoffwechselpraxis Bochum, Bochum, North Rhine-Westphalia
  - Private Practice - Dr. Claus Busch, Dr. Christian Busch & Dr. Christopher Cramer, Dortmund, North Rhine-Westphalia
  - InnoDiab Forschung Gmbh, Essen, North Rhine-Westphalia
  - Medizentrum Essen Borbeck, Essen, North Rhine-Westphalia
  - Private Practice - Dr. Bernd Becker, Essen, North Rhine-Westphalia
  - Institut für Diabetesforschung GmbH Münster, Münster, North Rhine-Westphalia
  - Diabetologikum Ludwigshafen/Die Praxis am Ludwigsplatz, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Diabetologische Schwerpunktpraxis Diabetologikum Speyer, Speyer, Rhineland-Palatinate
  - Practice Dr.med. Denger and Dr.med. Pfitzner, Friedrichsthal, Saarland
  - Zentrum für klinische Studien, Saint Ingbert, Saarland
  - Hausärztlich-Kardiologisches MVZ am Felsenkeller GmbH/Zentrum für klinische Studien, Dresden, Saxony
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden, Saxony
  - Velocity Clinical Research Leipzig GmbH, Leipzig, Saxony
  - Gemeinschaftspraxis Dr. Taeschner/Dr. Bonigut, Leipzig, Saxony
  - AmBeNet GmbH, Leipzig, Saxony
  - Private Practice - Dr. Christine Kosch, Pirna, Saxony
  - MVZ Riesa am Klinikum Döbeln GmbH, Riesa, Saxony
  - Praxis für Inner Medizin - Diabetologische Schwerpunktpraxis, Zwenkau, Saxony
  - Hausarzt- und Diabetologische Schwerpunktpraxis Hohenmölsen - Weiβenfels, Hohenmölsen, Saxony-Anhalt
  - SMO.MD GmbH, Magdeburg, Saxony-Anhalt
  - Universität zu Lübeck - Institut für Endokrinologie und Diabetes, Lübeck, Schleswig-Holstein
  - RED-Institut GmbH, Oldenburg in Holstein, Schleswig-Holstein
  - Private Practice - Dr. Joachim Weimer, Reinfeld, Schleswig-Holstein
  - Medizinisches Versorgungszentrum am Bahnhof Spandau, Spandau, State of Berlin
  - Gemeinschaftspraxis für Diabetologie, Eisenach, Thuringia
  - Institut für klinische Forschung und Entwicklung, Berlin
  - Diabetespraxis Prenzlauer Alle, Berlin
  - Diabetologische Schwerpunktpraxis Harburg, Hamburg
  - Diabetes Zentrum Wilhelmsburg, Hamburg
  - Diabeteszentrum Hamburg West, Hamburg
  - St. Josefskrankenhaus Heidelberg, Heidelberg
- Greece (10):
  - Athens Euroclinic, Athens, Attikí (Region)
  - Iatriko Paleou Falirou Medical Center, Palaió Fáliro, Attikí (Region)
  - General Hospital of Athens "G. Gennimatas", Athens, Attikí
  - Attikon General University Hospital, Chaïdári, Attikí
  - Ippokrateio General Hospital of Thessaloniki, Thessaloniki, Kentrikí Makedonía
  - Thermi Clinic, Thermi, Thessaloniki, Thessaloníki
  - AHEPA University General Hospital of Thessaloniki, Thessaloniki, Thessaloníki
  - Euromedica General Clinic of Thessaloniki, Thessaloniki, Thessaloníki
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki, Thessaloníki
  - University General Hospital of Larissa, Larissa, Thessalía
- Hungary (17):
  - Studium Egeszseghaz Kft, Kalocsa, Bács-Kiskun county
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged, Csongrád megye
  - Fejér Megyei Szent György Egyetemi Oktató Kórház, Székesfehérvár, Fejér
  - Debreceni Egyetem Kenézy Gyula Egyetemi Kórház, Debrecen, Hajdú-Bihar
  - Markhot Ferenc Oktatókórház, Eger, Heves County
  - Pharma 4 Trial, Gyöngyös, Heves County
  - Selye János Kórház, Komárom, Komárom-Esztergom
  - CLINFAN Szolgáltató Kft, Szekszárd, Tolna County
  - DRC Gyógyszervizsgáló Központ, Balatonfüred, Veszprém megye
  - Kanizsai Dorottya Korhaz, Nagykanizsa, Zala County
  - Zala Megyei Szent Rafael Kórház, Zalaegerszeg, Zala County
  - Szent Margit Rendelőintézet Nonprofit Kft, Budapest
  - ClinDiab Kft., Budapest
  - Szent János Kórház, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Strazsahegy Medicina Bt., Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
- India (14):
  - Gujarat Endocrin Pvt Ltd, Ahmedabad, Gujarat
  - Marengo CIMS Hospital, Ahmedabad, Gujarat
  - Bangalore Diabetes Centre, Bangalore, Karnataka
  - CARE CHL-Hospitals, Indore, Madhya Pradesh
  - Topiwala National Medical College & B. Y. L. Nair Charitable Hospital, Mumbai, Maharashtra
  - King Edward Memorial Hospital & Seth Gordhandas Sunderdas Medical College, Mumbai, Maharashtra
  - Kingsway Hospitals (Best Multispeciality Hospital in Nagpur), Nagpur, Maharashtra
  - G.B. Pant Institute of Postgraduate Medical Education & Research, New Delhi, National Capital Territory of Delhi
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Batra Hospital and Medical Research Centre, New Delhi, National Capital Territory of Delhi
  - Madras Diabetes Research Foundation, Chennai, Tamil Nadu
  - Care Hospitals Hyderabad- Banjara Hills, Hyderabad, Telangana
  - Apollo Multispeciality Hospitals limited, Kolkata, West Bengal
- Israel (23):
  - Edith Wolfson Medical Center, Holon, Central District
  - Meir Medical Center, Kfar Saba, Central District
  - Rabin Medical Center - Hasharon Campus, Petah Tikva, Central District
  - Rabin Medical Center, Petah Tikva, Central District
  - Sheba Medical Center, Ramat Gan, Central District
  - Kaplan Medical Center, Rehovot, Central District
  - Shaare Zedek Medical Center, Jerusalem, Jerusalem
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Hadassah Mount Scopus Medical Centre, Jerusalem, Jerusalem
  - Clalit Health Services Diabetes and Endocrinology Clinic Jerusalem, Jerusalem, Jerusalem
  - Emek Medical Center, Afula, Northern District
  - Hillel Yaffe Medical Center, Hadera, Northern District
  - Rambam Health Care Campus, Haifa, Northern District
  - Galilee Medical Center, Nahariya, Northern District
  - Holy Family Hospital, Nazareth, Northern District
  - ZIV Medical Center, Safed, Northern District
  - Clalit Health Services - Sakhnin Community Clinic, Sakhnin, Northern District
  - Barzilai Medical Center, Ashkelon, Southern District
  - Soroka Medical Center, Beersheba, Southern District
  - Sourasky Medical Center, Tel Aviv, Tell Abīb
  - Clalit Health Services - Atlit, Atlit, Ḥeifā
  - Bnai Zion Medical Center, Haifa, Ḥeifā
  - Linn Medical Center, Haifa, Ḥeifā
- Italy (20):
  - A.O.U.C. Policlinico di Bari, Bari, Apulia
  - Universita degli Studi della Campania Luigi Vanvitelli, Napoli, Campania
  - Fondazione Policlinico Tor Vergata, Rome, Lazio
  - Fondazione Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - Ospedale San Giovanni Calibita Fatebenefratelli, Rome, Lazio
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo, Lombardy
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Ospedale san Giovanni di Dio-Diabetologia, Olbia, Sardinia
  - A.O.U. Policlinico Paolo Giaccone, Palermo, Sicily
  - Ospedale Maggiore Pronto Soccorso, Chieri, Torino
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Azienda Ospedaliera Universitaria Pisana, Pisa, Tuscany
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Borgo Trento, Verona, Veneto
  - IRCCS - AOU di Bologna, Bologna
  - Azienda Ospedaliera Garibaldi, Catania
  - Azienda Ospedaliera Mater Domini, Catanzaro
  - Università degli Studi Gabriele D' Annunzio, Chieti
  - Centro Cardiologico Monzino, Milan
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Fondazione Salvatore Maugeri Clinica del lavoro, Pavia
- Japan (9):
  - Uji-Tokushukai Medical Center, Uji, Kyoto
  - Takatsuki Red Cross Hospital, Takatsuki, Osaka
  - The Institute of Medical Science, Asahi Life Foundation, Chuo-ku, Tokyo
  - Tokyo-Eki Center-building Clinic, Chuo-ku, Tokyo
  - Fukuwa Clinic, Chuo-ku, Tokyo
  - Medical Corporation Sato Medical clinic, Ootaku, Tokyo
  - Jinnouchi Hospital, Kumamoto
  - AMC Nishiumeda Clinic, Osaka
  - Sakurabashi Watanabe Advanced Healthcare Hospital, Osaka
- Mexico (24):
  - Centro de Investigacion Cardiovascular y Metabólica, Tijuana, Estado de Baja California
  - Diseno y Planeacion en Investigacion Medica, Guadalajara, Jalisco
  - Unidad de Investigaci�n Cl�nica Cardiometabolica de Occidente, Guadalajara, Jalisco
  - Centro de Investigacion Medica Integral, Guadalajara, Jalisco
  - Centro de Investigacion Medica de Occidente, S.C., Guadalajara, Jalisco
  - Universidad de Guadalajara, Guadalajara, Jalisco
  - Instituto Jalisciense de Investigacion en Diabetes y Obesidad, Guadalajara, Jalisco
  - Private Practice - Dr. Arechavaleta Granell Maria del Rosario, Guadalajara, Jalisco
  - Salud Cardiovascular, Guadalajara, Jalisco
  - Centro Especializado En Diabetes, Obesidad Y Prevencion De Enfermedades Cardiovasculares, Mexico City, Mexico City
  - Instituto de Diabetes, Obesidad y Nutricion, Cuernavaca, Morelos
  - Cardiolink Clin Trials, Monterrey, Nuevo León
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - Unidad Médica para la Salud Integral, San Nicolás de los Garza, Nuevo León
  - Centro Para El Desarrollo de La Medicina Y de Asistencia Medica Especializada S.C., Culiacán, Sinaloa
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares, Ciudad Madero, Tamaulipas
  - Hospital Angeles Xalapa, Xalapa, Veracruz
  - Medical Care and Research SA de CV, Mérida, Yucatán
  - Centro de Investigacion Medica Aguascalientes, Aguascalientes
  - Fundación Cardiovascular de Aguascalientes A.C., Aguascalientes
  - Hospital Cardiologica Aguescalientes, Aguascalientes
  - Investigacion En Salud Y Metabolismo S.C / Nutricion Clinica / Unidad de Base de Datos, Chihuahua City
  - Lahoja. Asociacion Para La Investigacion Y La Farmacovigilancia, Durango
  - Centro de Estudios Clínicos de Querétaro (CECLIQ), Querétaro
- Netherlands (18):
  - Ziekenhuis Bethesda, Hoogeveen, Drenthe
  - EB Utrecht, Almere Stad, Flevoland
  - Ziekenhuis Rijnstate, Arnhem, Gelderland
  - Slingeland Ziekenhuis, Doetinchem, Gelderland
  - Ziekenhuis Gelderse Vallei, Ede, Gelderland
  - Radboudumc, Nijmegen, Gelderland
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen, Gelderland
  - Jeroen Bosch ziekenhuis, 's-Hertogenbosch, North Brabant
  - Ziekenhuis Amstelland, Amstelveen, North Holland
  - Amsterdam UMC, locatie VUmc, Amsterdam, North Holland
  - Amsterdam UMC, locatie AMC, Amsterdam, North Holland
  - Spaarne Gasthuis, Haarlem Zuid, Haarlem, North Holland
  - Saxenburgh Medisch Centrum, Hardenberg, Overijssel
  - Reinier de Graaf Ziekenhuis, locatie Delft, Delft, South Holland
  - Het Van Weel-Bethesda Ziekenhuis - Ziekenhuis Dirksland, Dirksland, South Holland
  - Franciscus Gasthuis & Vlietland, Locatie Gasthuis, Rotterdam, South Holland
  - Diakonessenhuis, locatie Utrecht, Utrecht
  - Universitair Medisch Centrum Utrecht, Utrecht
- Poland (19):
  - OMEDICA Medical Center, Poznan, Greater Poland Voivodeship
  - Gaja Poradnie Lekarskie Maciej Wiza, Poznan, Greater Poland Voivodeship
  - Private Practice - Dr. Ewa Krzyzagorska, Poznan, Greater Poland Voivodeship
  - Medyczne Centrum Diabetologiczno Endokrynologiczno Metaboliczne DIAB-ENDO-MET, Krakow, Lesser Poland Voivodeship
  - Private Practice - Dr. Robert Witek, Tarnów, Lesser Poland Voivodeship
  - NZOZ Regionalna Poradnia Diabetologiczna, Wroclaw, Lower Silesian Voivodeship
  - Wojewódzki Zespól Specjalistycznej Opieki Zdrowotnej, Wroclaw, Lower Silesian Voivodeship
  - CenterMed Lublin NZOZ, Lublin, Lublin Voivodeship
  - Gabinety TERPA, Lublin, Lublin Voivodeship
  - NZOZ Medica, Lublin, Lublin Voivodeship
  - Centrum Medyczne AMED, Warsaw, Masovian Voivodeship
  - Instytut Diabetologii, Warsaw, Masovian Voivodeship
  - ETG NETWORK Sp. z o.o., Warsaw, Masovian Voivodeship
  - Legeartis - Poradnie Specjalistyczne, Bialystok, Podlaskie Voivodeship
  - Niepubliczny Specjalistyczny Zaklad Opieki Zdrowotnej Osrodek Diabetologiczny Popula Spolka Cywilna, Bialystok, Podlaskie Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk, Pomeranian Voivodeship
  - NZOZ Salvia CM, Katowice, Silesian Voivodeship
  - NZOZ Przychodnia Specjalistyczna Andrzej Wittek, Henryk Rudzki, Ruda Śląska, Silesian Voivodeship
  - Centrum Terapii Wspolczesnej J. M. Jasnorzewska Spolka Komandytowo-Akcyjna, Lodz, Łódź Voivodeship
- Puerto Rico (5):
  - Advanced Clinical Research, LLC, Bayamón
  - Manati Center for Clinical Research, Manatí
  - Research and Cardiovascular Corp., Ponce
  - GCM Medical Group, PSC - Hato Rey Site, San Juan
  - San Juan City Hospital, San Juan
- Romania (20):
  - Private Practice - Dr. Diana Barbonta, Alba Iulia, Alba
  - Diabdana, Oradea, Bihor County
  - Centrul Medical Grandmed, Oradea, Bihor County
  - C.M.D.T.A. Neomed, Brasov, Brașov County
  - Nicodiab, Bucharest, București
  - Geea Medical Easy Diet, Bucharest, București
  - Centrul Medical NutriLife, Bucharest, București
  - The National Institute of Diabetes, Nutrition and Metabolic Diseases "Prof. Dr. N. Paulescu", Bucharest, București
  - Gama Diamed, Mangalia, Constanța County
  - Top Diabet SRL, Craiova, Dolj
  - CMI DNBM Dr. Pop Lavinia, Baia Mare, Maramureş
  - SC Dentosim Queen SRL - Centrul Medical Diamed, Târgu Mureş, Mureș County
  - Diabmed Dr. Popescu Alexandrina, Ploieşti, Prahova
  - Dianutrilife Medica, Ploieşti, Prahova
  - Centru Medical Dr. Negrisanu, Timișoara, Timiș County
  - CMI Dr.Pletea Noemi SRL, Bacau
  - SC Minimed SRL, Bacau
  - Diamed Obesity, Galați
  - Olimpia Med, Iași
  - Centrul Medical Consultmed, Iași
- Russia (22):
  - Arkhangelsk Regional Clinical Hospital, Arkhangelsk, Arkhangelskaya oblast
  - First City Clinical Hospital E.E. Volosevich, Arkhangelsk, Arkhangelskaya oblast
  - Advisory Diagnostic Centre, Syktyvkar, Komi
  - City Mariinskaya Hospital, Saint Petersburg, Leningradskaya Oblast'
  - National Medical Research Center for therapy and preventive medicine, Moscow, Moscow
  - Endocrinology Research Center of Rosmedtechnologies, Moscow, Moscow
  - Pirogov Russian National Research Medical University, Moscow, Moscow
  - First Moscow State Medical University I.M. Sechenov, Moscow, Moscow
  - Russian Cardiology Research and Production Complex, Moscow, Moscow
  - Moscow City Clinical Hospital Number 52, Moscow, Moscow
  - M. F. Vladimirskiy Moscow Regional Research Clinical Institute, Moscow, Moscow
  - Novosibirsk State Medical University, Novosibirsk, Novosibirsk Oblast
  - Rostov State Medical University, Rostov-on-Don, Rostov Oblast
  - Ryazan Regional Clinical Cardiological Dispensary, Ryazan, Ryazan Oblast
  - S.M. Kirov Military Medical Academy, Saint Petersburg, Sankt-Peterburg
  - Saint-Petersburg City Hospital of Saint Elizabeth, Saint Petersburg, Sankt-Peterburg
  - Astarta Clinic, Saint Petersburg, Sankt-Peterburg
  - Regional Clinical Hospital of the Saratov Region, Saratov, Saratov Oblast
  - Tomsk Regional Clinical Hospital, Tomsk, Tomsk Oblast
  - Siberian State Medical University, Tomsk, Tomsk Oblast
  - Research & Practice, Yaroslavl, Yaroslavl Oblast
  - Yaroslavl State Med Acad Clinical Hospital, Yaroslavl, Yaroslavl Oblast
- Slovakia (9):
  - IN-DIA, Lučenec, Banská Bystrica Region
  - Diacrin s.r.o., Bratislava, Bratislava Region
  - Sin Azucar, Malacky, Bratislava Region
  - DIAB sro, Rožňava, Košice Region
  - Funkystuff, Nové Zámky, Nitra Region
  - Diabetol, Prešov, Presov
  - MED-DIA s.r.o, Sabinov, Presov
  - DIA-MED CENTRUM s.r.o., Púchov, Trenčín Region
  - Diabetes Centrum, Trenčín, Trenčín Region
- South Korea (10):
  - Yonsei University-Wonju Severance Christian Hospital, Wŏnju, Kang-won-do
  - Korea University Anam Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [Seoul]
  - Kyung Hee University Hospital at Gangdong, Seoul, Seoul-teukbyeolsi [Seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Hallym University Kangnam Sacred Heart Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Keimyung University Dongsan Hospital, Daegu, Taegu-Kwangyǒkshi
  - Ulsan University Hospital, Ulsan, Ulsan-Kwangyǒkshi
- Spain (20):
  - CHUAC-Complejo Hospitalario Universitario A Coruña, A Coruña, A Coruña [La Coruña]
  - Complejo Hospitalario Universitario de Ferrol (CHUF)- Hospital Naval, Ferrol, A Coruña [La Coruña]
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela, A Coruña [La Coruña]
  - Centro Periférico de Especialidades Bola Azul, Almería, Almería
  - Hospital Universitario Virgen de la Victoria, Málaga, Andalusia
  - Hospital Quiron Infanta Luisa, Seville, Andalusia
  - Hospital Universitario Central de Asturias, Oviedo, Asturias, Principado de
  - Hospital Clínico Universitario de Valladolid, Valladolid, Castille and León
  - Hospital Virgen del Camino, Sanlúcar de Barrameda, Cádiz
  - Hospital Virgen de las Montañas, Villamartín, Cádiz
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Príncipe de Asturias, Alcalá de Henares, Madrid, Comunidad de
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Comunidad de
  - Hospital General Universitario de Valencia, Valencia, Valenciana, Comunitat
  - Hospital Universitario de La Ribera, Alzira, València
  - Hospital Unviersitario Virgen Nieves, Granada
  - Hospital Universitario La Paz, Madrid
  - Clínica nuevas Tecnologías en Diabetes y Endocrinología (NTDE), Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sweden (6):
  - Dalecarlia Clinical Research Center, Rättvik, Dalarnas Län [se-20]
  - Östersunds Sjukhus, Östersund, Jämtlands Län [se-23]
  - ProbarE, Lund, Skåne Län [se-12]
  - Citydiabetes, Stockholm, Stockholms Län [se-01]
  - Sahlgrenska Universitetssjukhuset Mölndal, Mölndal, Västra Götalands Län [se-14]
  - Universitetssjukhuset Örebro, Örebro, Örebro Län [se-18]
- Taiwan (9):
  - Changhua Christian Hospital, Changhua County, Changhua
  - Mackay Memorial Hospital-Hsinchu, Hsinchu, Hsinchu
  - Hualien Tzu Chi Medical Center, Hualien City, Hualien
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist, Kaohsiung
  - Chi Mei Medical Center, Tainan, Tainan
  - Taichung Veterans General Hospital, Taichung
  - National Cheng-Kung Uni. Hosp., Tainan
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- Turkey (Türkiye) (19):
  - Baskent University Dr. Turgut Noyan Research and Training Center, Yüreğir, Adana
  - Dicle Üniversitesi, Sur, Diyarbakır
  - Eskisehir Osmangazi University, Eskişehir, Eskişehir
  - Dokuz Eylül Üniversitesi, Balçova, İzmir
  - Ege Universitesi Hastanesi, Bornova, İzmir
  - Mersin University Medical Faculty, Yenişehir, Mersin
  - Akdeniz Universitesi Hastanesi, Antalya
  - Adnan Menderes University Medical Faculty, Aydin
  - Pamukkale University Medical Faculty, Fahri Goksin Oncology Centre, Denizli
  - Atatürk Üniversitesi, Erzurum
  - Gaziantep Üniversitesi Gaziantep Onkoloji Hastanesi, Gaziantep
  - Koç Üniversitesi Hastanesi, Istanbul
  - Dr. Sadi Konuk Egitim ve Arastirma Hastanesi, Istanbul
  - Acibadem Universitesi Atakent Hastanesi, Istanbul
  - Göztepe Eitim Ve Aratrma Hastanesi, Istanbul
  - Fatih Sultan Mehmet Training and Research Hospital, Istanbul
  - Erciyes University Medical Faculty, Kayseri
  - Kocaeli Üniversitesi, Kocaeli
  - İnönü Üniversitesi Turgut Özal Tıp Merkezi, Malatya
- Ukraine (20):
  - Regional Communal Non-commercial enterprise "Chernivtsi regional clinical hospital", Chernivtsi, Chernivetska Oblast
  - Dnipropetrovsk City Clinical Hospital No. 9, Dnipro, Dnipropetrovsk Oblast
  - Ukrainian State Research Institute Of Medical And Social Problems Of Disability, Dnipro, Dnipropetrovsk Oblast
  - City Clinical Hospital No. 2, Kharkiv, Kharkivs’ka Oblast’
  - L.T. Mala National Institute of Therapy of NAMS of Ukraine, Kharkiv, Kharkivs’ka Oblast’
  - Municipal Non-Profit Enterprise "City clinical hospital №8" of Kharkiv city council, Kharkiv, Kharkivs’ka Oblast’
  - Institute of Endocrinology and Metabolism named after Komissarenko, Kiev, Kyiv Oblast
  - Medical Center of Limited Liability Company "Medical Center "Consilium Medical", Kiev, Kyiv Oblast
  - ARTEM, Kiev, Kyivska Oblast
  - Medbud Clinic, Kyiv, Kyivska Oblast
  - Branch "Center of Endocrinological Health" of "Lviv Regional Clinical Diagnostic Center", Lviv, Lviv Oblast
  - Lviv City Clinical Hospital #4, Lviv, Lviv Oblast
  - Municipal non-profit enterprise'Odesa Regional Clinical Hospital'of Odesa Regional Council, Odesa, Odesa Oblast
  - Municipal non-profit enterprise "Consultative-diagnostic center №20" of Odesa city council, Odesa, Odesa Oblast
  - Poltova Oblast Clinical Hospital IM.M.V.Sklifosovskoho, Poltava, Poltava Oblast
  - Municipal enterprise "1st City clinical hospital of Poltava City Council", Poltava State Medical University, Poltava, Poltava Oblast
  - Municipal Non-Profit Enterprise Of Sumy Regional Council ''Sumy Regional Clinical Hospital'', Sumy, Sumska Oblast
  - Vinnytsia Regional Clinical Endocrinology Dispensary, Vinnytsia, Vinnytsia Oblast
  - Municipal non-profit enterprise "City Hospital #7" of Zaporizhzhia City Council, Zaporizhzhya, Zaporizhzhia Oblast
  - Medical Center Ok!Clinic+, Kyiv
- United Kingdom (12):
  - Aberdeen Royal Infirmary, Aberdeen, Aberdeen City
  - Ninewells Hospital and Medical School, Dundee, Angus
  - Southmead Hospital, Bristol, Bristol, City of
  - Staploe Medical Centre, Ely, Cambridgeshire
  - Knowle House Surgery, Plymouth, Devon
  - The Royal Cornwall Hospital, Truro, England
  - Glasgow Royal Infirmary, Glasgow, Glasgow City
  - Hull Royal Infirmary, Hull, Kingston Upon Hull
  - Leicester General Hospital, Leicester, Leicestershire
  - Ipswich Hospital, Ipswich, Suffolk
  - Morriston Hospital, Swansea, Swansea [Abertawe Gb-ata]
  - University Hospital Aintree, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Nicholls SJ, Pavo I, Bhatt DL, Buse JB, Del Prato S, Kahn SE, Lincoff AM, McGuire DK, Miller D, Nauck MA, Nishiyama H, Nissen SE, Sattar N, Weerakkody G, Wiese RJ, Zinman B, Zoungas S, Basile J, Davies MJ, Giorgino F, Kellerer M, Ji L, Varkonyi T, Menon V, Broder JC, Herschtal A, D'Alessio D; SURPASS-CVOT Investigators. Cardiovascular Outcomes with Tirzepatide versus Dulaglutide in Type 2 Diabetes. N Engl J Med. 2025 Dec 18;393(24):2409-2420. doi: 10.1056/NEJMoa2505928. PMID 41406444
- [Derived] Khawaji A, A Jaly A, A Bakri H, Ravi R, Hattan A, Khawaji A, Najmi W. Weight Loss Efficacy of Tirzepatide Compared to Placebo or GLP-1 Receptor Agonists in Adults With Obesity or Overweight: A Meta-Analysis of Randomized Controlled Trials With >/= 20 Weeks Treatment Duration. J Obes. 2025 Jul 24;2025:3442754. doi: 10.1155/jobe/3442754. eCollection 2025. PMID 40746703
- [Derived] Kaneko S. Tirzepatide: A Novel, Once-weekly Dual GIP and GLP-1 Receptor Agonist for the Treatment of Type 2 Diabetes. touchREV Endocrinol. 2022 Jun;18(1):10-19. doi: 10.17925/EE.2022.18.1.10. Epub 2022 Jun 16. PMID 35949358
- See also: A Study of Tirzepatide (LY3298176) Compared With Dulaglutide on Major Cardiovascular Events in Participants With Type 2 Diabetes — https://trials.lillytrialguide.com/en-US/trial/7Hobv37NARjOCQyknTYfRZ